CLINICAL TRIAL: NCT06038123
Title: China CIED 3.0T MRI Performance Study
Brief Title: China 3T MRI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT23009
Record Dates: First submitted 2023-09-05; First posted 2023-09-14 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2024-10

CONDITIONS: Bradycardia; Tachycardia; Heart Failure
MeSH Terms: conditions — Bradycardia; Tachycardia; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with market released 3.0T conditional CIED systems undergoing 3.0T MRI scan attempt (Experimental): This was a single-arm study to confirm safety and effectiveness of the SureScan CIED System in the clinical MRI environment when subjects receive 3.0T MRI scans without positioning restrictions (MRI scans may occur anywhere on the body). Study devices refer to China market released 3.0T Magnetic resonance (MR) conditional CIED systems. Subjects implanted with a SureScan study device who underwent a 3.0T MRI scan attempt were considered in endpoint analyses.
  Interventions: Device: China market released 3.0T Magnetic resonance (MR) conditional CIED systems

INTERVENTIONS:
Device: China market released 3.0T Magnetic resonance (MR) conditional CIED systems — To confirm safety and effectiveness of the SureScan CIED System in the clinical MRI environment when subjects receive 3.0T MRI scans without positioning restrictions (MRI scans may occur anywhere on the body)

SUMMARY:
The purpose of the China CIED 3.0T MRI Performance Study is to confirm safety of SureScan CIED in the clinical 3.0T MRI environment when subjects receive MRI scans. All subjects will have required follow-up visits at baseline, MRI visit, 1-month post-MRI. The MRI scans will occur at the MRI visit. The MRI scan region will be determined by investigator according to the subject's clinical condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were implanted an SureScan system CIED over 6 weeks at the time of signing ICF.
* Subjects who are able and willing to undergo elective MRI scanning without sedation.
* Subjects who were implanted an SureScan system CIED in the pectoral region.
* Subjects who are geographically stable and available for follow-up at the study site for the length of the study.
* Subjects who are at least 18 years of age (or older, if required by local law).

Exclusion Criteria:

* Subjects who require a legally authorized representative to obtain informed consent.
* Subjects with abandoned or capped leads.
* Subjects who require an indicated MRI scan, other than those specifically described in the China CIED 3.0T MRI performance study, before the 1-month post-MRI follow-up.
* Subjects with a non-MRI compatible device (such as neurostimulators) or material implant (e.g., non-MRI compatible sternal wires, neurostimulators, biostimulators, metals or alloys).
* Subjects with medical conditions that preclude the testing required by the CIP or limit study participation.
* Subjects who are enrolled or intend to participate in another clinical trial (of an investigational drug or device, new indication for an approved drug or device, or requirement of additional testing beyond standard clinical practice) during the SureScan study. Co-enrollment in concurrent trials is only allowed when documented pre-approval is obtained from the Medtronic study manager.
* Female patient who is pregnant, or of childbearing potential and not on a reliable form of birth control. Women of childbearing potential are required to have a negative pregnancy test within seven (7) days prior to device implant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Shanghai Tongren Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first site was activated on 27 Nov 2023 and the first subject was enrolled on 28 November 2023. The last subject enrollment occurred on 27 August 2024. Sites were notified of enrollment completion on 27 Aug 2024. Sites were instructed to exit subjects starting 17 Oct 2024 to close the study. The last study exit occurred on 28 October 2024. Overall, 64 subjects enrolled at 5 clinical sites in mainland China.
Pre-assignment Details: Among the 64 enrolled subjects, 1 subject exited the study without having an MRI attempt and 63 subjects underwent an MRI attempt. Of the 63 subjects who had an MRI attempt, 61 completed the 1-month post MRI visit and exited the study afterwards because of study completion, and the other 2 subjects missed the 1-month post MRI visit due to subject withdrawal (1) and femur fracture (1).
Period: Overall Study
Arm/Group | Subjects With Market Released 3.0T Conditional CIED Systems Undergoing 3.0T MRI Scan Attempt
Started | 63
Completed | 61
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — not return due to femur fracture | 1

BASELINE CHARACTERISTICS:
Population: Among the 64 enrolled subjects, one subject exited the study before an MRI attempt due to withdrawal by subject; this subject did not have baseline information collected. Therefore, baseline characteristics summarized for the 63 subjects who underwent a 3.0T MRI scan attempt.
Arm/Group | Subjects With Market Released 3.0T Conditional CIED Systems Undergoing 3.0T MRI Scan Attempt
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
New York Heart Association (NYHA) Classification [Count of Participants; unit: Participants]
  Class I (Mild): No symptoms with ordinary physical activity; no limitation of activity. | 2
  Class II (Mild): Slight limitation of activity | 21
  Class III (Moderate): Marked limitation of activity | 15
  Class IV (Severe): Inability to carry on any physical activity without discomfort | 0
  Subject does not have heart failure | 25

OUTCOME MEASURES:

1. Primary Outcome: The Occurrence of an MRI-related Event for CIED
Description: The primary objective was to demonstrate the safety of SureScan system CIED in clinical 3.0T MRI environment within 1-month post-MRI scan. Specifically, it was hypothesized that the MRI-related event-free rate within 1-month post-MRI to be greater than 90%. The proportion of subjects free from MRI-related events was calculated by dividing the number of subjects without an MRI-related event by the number of subjects at risk for an event. The occurrence of any of the following within 30 days after a 3.0T MRI scan would be considered an MRI-related event: (1) Medical advisor-assessed MRI-related complication within 30 days post-MRI (for iPG, ICD or CRT-D); (2) Medical advisor-assessed right ventricular MRI-related loss of capture within 30 days post-MRI (for iPG, ICD or CRT-D); (3) Sustained tachyarrhythmia originating during SureScan programming, requiring immediate treatment (defined as ATP, device shock, or external shock), as assessed by a medical advisor (for ICD or CRT-D).
Time Frame: The event will be collected within 30 days after MRI visit.
Population: Of the 63 patients who underwent an MRI attempt, 4 patients were not qualified for the analysis (including 2 patients for whom device testing was not done at both pre- and post-MRI visits, 1 patient who did not meet pre-MRI requirements and missed 1-month post MRI visit, and 1 patient who missed 1-month post MRI visit). The remaining 59 patients were included in the endpoint analysis for MRI-related events.
Measure: Count of Participants; unit: Participants
Groups:
- Subjects With a SureScan Study Device Completing 3.0T MRI Scan and 1-month Post MRI Follow-up Visit: All subjects implanted with a SureScan study device who have a 3.0T MRI scan after enrollment and have completed their one-month post-MRI scan follow-up, or have had an MRI-related event without completion of their one-month post-MRI scan follow-up will be included in the main analysis for the primary objective.
Arm/Group | Subjects With a SureScan Study Device Completing 3.0T MRI Scan and 1-month Post MRI Follow-up Visit
Number analyzed (Participants) | 59
Participants
  Without MRI-related events within 1-month post MRI visit | 59
  With MRI-related events within 1-month post MRI | 0
Statistical Analysis 1: Comparison: Subjects With a SureScan Study Device Completing 3.0T MRI Scan and 1-month Post MRI Follow-up Visit; Alternative hypothesis: MRI-related event-free rate within 1-month post-MRI >90%. Null hypothesis will be rejected if the one-sided 97.5% lower confidence bound is >90%. Assuming type I error rate of 0.025, even-free rate under null hypothesis being 90% and true even-free rate being 99.5%, the minimum required sample size is 54 MRI scanned patients to achieve 90% power. One-proportion binomial exact test along with a one-sided 97.5% lower (Clopper-Pearson) confidence bound was used; Test type: Superiority; p = 0.002, One-proportion binomial exact test — A priori threshold for statistical significance was 0.025; Proportion = 100, 97.5% CI 1-sided [lower limit 93.94]

2. Secondary Outcome: The Changes in Atrial and Ventricular Pacing Capture Thresholds From Pre-MRI to 1-month Post-MRI Scan.
Description: There was no hypothesis for this secondary objective. Pacing capture thresholds (PCTs) to be characterized include:
  APCT of atrial lead for subjects with an IPG device; APCT of atrial lead and VPCT of right ventricular (RV) lead for subjects with an ICD device; APCT of atrial lead and VPCTs of right ventricular (RV) and left ventricular (LV) leads for those with a CRT-D device.
  PCTs of each subject will be measured prior to the 3.0T MRI scan and at the one-month post-MRI. Change in PCT is defined as PCT measured at one-month post-MRI subtracts that measured prior to a 3.0T MRI scan. Proportion of subjects with an increase less than or equal to 0.5V in APCT or VPCTs from pre-MRI to one-month post-MRI will also be used to characterize the efficacy performance of SureScan with respect to PCTs. If the 1-month post-MRI APCT or VPCT is missing, the PCT measured immediately post-MRI will be used instead.
Time Frame: The evaluation will be compared from pre-MRI to 1-month post-MRI scan
Population: The following changes in PCTs were evaluated using descriptive statistics:
  * Right atrial lead measured in 45 patients, attrition: device testing not done (2) , no exiting lead (11), unable to lose capture (1), pre-MRI requirements not met/missing (4).
  * Right ventricular lead measured in 60 patients, attrition: device testing not done (2), pre-MRI requirements not met (1).
  * Left ventricular lead measured in 9 patients, attrition: device testing not done (2), no existing lead (n=52).
Measure: Mean (Standard Deviation); unit: Volt
Groups:
- Subjects With a SureScan Study Device Undergoing a 3.0T MRI Scan Attempt: To be included in the analysis for pacing capture thresholds (PCTs), all the following must be met:
  1. The subject must undergo a 3.0T MRI scan.
  2. The subject must have valid PCT measurements pre- and post-MRI (see paragraph below for definitions).
  3. The (atrial, right or left ventricular) lead is not dislodged within 6 weeks prior to MRI scan.
  4. The (atrial, right or left ventricular) lead has not been replaced or repositioned within 6 weeks prior to MRI scan or between MRI scan and the one-month post-MRI visit.
  5. The VPCTs of RV at the pre-MRI must be ≤ 2.0V. This is because subjects with a higher VPCT cannot have an MRI per CIP
  To be a valid PCT measurement, the pulse width must be set to 0.4ms and a printed pacing capture threshold testing strip must be available to confirm the pulse width and capture threshold reported. The pre-MRI period value will be the pre-MRI period PCT measurement. For the post-MRI period PCT value, the PCT value on the one-month post-MRI period CRF will be used. If that does not exist or is not valid, the PCT measured immediately post-MRI will be used instead.
Arm/Group | Subjects With a SureScan Study Device Undergoing a 3.0T MRI Scan Attempt
Number analyzed (Participants) | 63
Volt
  Change in PCT of right atrial lead: number analyzed (Participants) | 45
  Change in PCT of right atrial lead | -0.04 (0.17)
  Change in PCT of right ventricular lead: number analyzed (Participants) | 60
  Change in PCT of right ventricular lead | 0.02 (0.20)
  Change in PCT of left ventricular lead: number analyzed (Participants) | 9
  Change in PCT of left ventricular lead | 0.14 (0.42)

ADVERSE EVENTS:
Time Frame: Adverse events of all the 64 enrolled subjects were collected from enrollment to exit over an average of 178 days of follow-up.
Description: All adverse events (AEs) were collected throughout the study duration, starting at the time the Informed Consent Form was signed. Reporting of these events to Medtronic occurred on an AE form. Each event must be reported separately. Documented pre-existing conditions were not considered as reportable AEs unless the nature or severity of the condition had worsened.
Groups:
- Enrolled Subjects: All subjects enrolled in the study
Arm/Group | Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 5/64
Other Adverse Events (participants affected / at risk) | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=64)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, contracts allow investigators to publish study results per the protocol and publication plan. Investigators and participating institutions will provide any publication of study data generated by the Investigator and/or participating institution to Medtronic for review prior to submission to determine if confidential information ("CI") is included and to check for technical correctness. Medtronic may not censor/interfere with the publication beyond the extent necessary to protect CI.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT06038123/Prot_SAP_000.pdf